CLINICAL TRIAL: NCT04297384
Title: Breast Cancer Pathways Impact on Patient Shared Decision Making and Experience in Academic and Community Practice
Brief Title: Breast Cancer Pathways Program Impact on Patient Shared Decision Making and Experience in Academic and Community Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I 60517; NCI-2019-07900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 60517 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Breast Carcinoma; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (standard educational materials, surveys) (Active Comparator): Participants receive standard chemotherapy educational materials. Participants also complete surveys over approximately 22 minutes at the time of first chemotherapy infusion, and approximately 8 weeks after first chemotherapy infusion.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration
- Group II (personalized information, surveys) (Experimental): Participants receive personalized information about their cancer, treatment, and side effects. Participants also complete surveys over approximately 22 minutes at the time of first chemotherapy infusion, and approximately 8 weeks after first chemotherapy infusion.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive standard chemotherapy educational materials
  Arms: Group I (standard educational materials, surveys)
Other: Informational Intervention — Receive personalized information about cancer, treatment, and side effects
  Arms: Group II (personalized information, surveys)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete surveys

SUMMARY:
This trial studies the impact of the breast cancer pathways program on the patient experience, including decision making and quality of life. Measuring how the breast cancer pathways program affects decision making and quality of life in patients may help doctors improve cancer education.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the impact of breast cancer pathways on patient experience, burden of decision making and quality of life in tertiary cancer center and community oncology practice.

II. Identify modifiable factors that affect provider adoption of breast cancer pathways in tertiary cancer center and community oncology practice.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Participants receive standard chemotherapy educational materials. Participants also complete surveys over approximately 22 minutes at the time of first chemotherapy infusion, and approximately 8 weeks after first chemotherapy infusion.

GROUP II: Participants receive personalized information about their cancer, treatment, and side effects. Participants also complete surveys over approximately 22 minutes at the time of first chemotherapy infusion, and approximately 8 weeks after first chemotherapy infusion.

ELIGIBILITY:
Inclusion Criteria:

* Treatment includes intravenous chemotherapy for breast cancer for primary disease as neoadjuvant or adjuvant therapy, or for recurrent and/or metastatic cancer
* Can provide consent
* Are able to comprehend written materials in English or Spanish
* Will receive their chemotherapy at Roswell Park sites in Buffalo or Amherst, New York (NY), or Roswell Park Oncology primary care (PC) sites in Niagara Falls, Amherst, West Seneca, or Jamestown NY

Exclusion Criteria:

* Breast cancer patients receiving oral therapy alone
* Patients who are not able to comprehend written materials in English or Spanish
* Patients who will not receive chemotherapy at a Roswell Park site
* Patients who are not able to comprehend written materials will not be included in this study, as the consent document will be administered in multiple infusion centers that cannot be all staffed daily with a research associate. The study instruments used are standardized tools that have been developed as best as possible with appropriate literacy levels
* Patients enrolled in clinical trials for their breast chemotherapy will be excluded from this study because they will require alternative educational materials that are specific to the trial drugs being administered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
change in Patient quality of life | Baseline and 8 weeks
  Assessed by surveys.
Change in Patient quality of decision | Baseline and 8 weeks
  Assessed by surveys
Number of physician visits and diagnostic tests | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Edge, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States